CLINICAL TRIAL: NCT06145542
Title: Sequences of Aerobic and Resistance Exercise in Training and Their Effects on Cardio-metabolic Functions Among Type 2 Diabetes Patients - a Randomized Study
Brief Title: Sequences of Aerobic and Resistance Exercise and Cardio-metabolic Functions in T2D
Acronym: ARRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Nanjing Sport Institute (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Xiao Tan, Associate Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RT-2023-17
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: aerobic exercise; resistance exercise; exercise order; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR group (Experimental): aerobic exercise then resistance exercise in all training sessions
  Interventions: Behavioral: AR group: aerobic training before resistance training
- RA group (Active Comparator): resistance exercise then aerobic exercise in all training sessions
  Interventions: Behavioral: RA group: resistance exercise before aerobic exercise

INTERVENTIONS:
Behavioral: AR group: aerobic training before resistance training — Exercise are performed 3 times/wk for 8 wks.
  Aerobic training sessions are performed using cycle ergometers. Riding speed is 55-60 rotations/min, at an intensity between 50%-75% of heart rate reserve (HRR). Real-time heart rate monitors are worn by each participant during the session. Aerobic training session lasts for 30 minutes, with an additional 5-minute warm-up and 5-min relaxation training before and after the session, respectively.
  Participants perform resistance exercise on a set of strength training equipment. Load of resistance exercise is between 60-80% of repetition maximum (RM) in each set of exercise. Six different groups of resistance exercise (involving contractions and relaxations of biceps, triceps, pectoralis major, latissimus dorsi, quadriceps, and hamstrings) are conducted, with 6 sets of 10 repeated tasks in each group. Participants are instructed to finish each set of exercise task within 60 seconds. Between each two sets, there are 60 s of rest time.
  Arms: AR group
Behavioral: RA group: resistance exercise before aerobic exercise — Exercise are performed 3 times/wk for 8 wks.
  Following a 5-min warm-up exercise, the participants perform resistance training on a set of equipment. Load of resistance exercise is set between 60-80% of repetition maximum in each set of exercise. Six different groups of resistance exercise (involving contractions and relaxations of biceps, triceps, pectoralis major, latissimus dorsi, quadriceps, and hamstrings) are conducted, with 6 sets of 10 repeated tasks in each group. Participants are instructed to finish each set of exercise task within 60 s. Between each two sets, there are 60 seconds of rest time.
  Aerobic training sessions are performed using cycle ergometers. Riding speed is 55-60 rotations/min, at an intensity between 50%-75% of heart rate reserve. Real-time heart rate monitors are worn during the entire session. Each aerobic training session lasts for 30 minutes, with an 5-minute relaxation training after the session.
  Arms: RA group

SUMMARY:
Aerobic exercise and resistance exercise are two types of exercise commonly used in physical conditioning. Compared to aerobic exercise, a combination of aerobic and resistance exercise has been linked to a greater reduction in hemoglobin A1c (HbA1c) among patients with type 2 diabetes (T2D). However, it is not clear that in a concurrent aerobic-resistance training session, whether the orders of the two types of exercise could act differently in glucose metabolism. This randomized trial aims to investigate the effect of the sequence of exercise modalities (aerobic-resistance vs resistance-aerobic in a training session) on glycemic control among T2D patients following an 8-wk intervention period.

DETAILED DESCRIPTION:
Objectives:

This randomized study aims to explore the effects of aerobic and resistance training sequences on glycemic control among type 2 diabetes (T2D) patients through an 8-wk combined aerobic and resistance exercise training program.

Study Population:

A total of 56 participants with T2D aged 50-70 years (sex ratio approximately 1:1) with a course of type 2 diabetes of more than one year are included. Participants are residents of Nanjing Municipality, Jiangsu Province, China. Participants are recruited from the outpatients at Maigaoqiao Community Health Service Center, Qixia District, Nanjing, China or through online advertisement published on the official social media (WeChat) channels of the Health Service Center.

Randomization:

Participants are stratified by baseline hemoglobin A1c (HbA1c) and age, they are randomly assigned into two groups with a block size of 4. The study groups are: 1) aerobic before resistance training (AR group, n=28); 2) resistance before aerobic training (RA group, n=28).

Exercises intervention program:

Exercised program is designed to take place three times a week for a total of eight weeks. Exercise intervention is scheduled for approximately 70 minutes per session (30 minutes of aerobic and 30 minutes of resistance, no break between two types, 5-min of preparation and 5-min relaxation stretching movements before and after each intervention), performed between 8:00 to 11:00 or between 14:00 to 16:30, Monday through Saturday.

Target heart rate during aerobic exercise is set as resting heart rate (HR) + 40%-70% of heart rate reserve (HRR). Participants' HRR was calculated based on their resting HR and maximum heart rate (HRmax=208-0.7×age) as HRmax - HR. Heart rate monitors (OH1, Polar Oy, Oulu, Finland) are used during all exercise sessions to track exercise intensity and ensure that it remained within the specified range. Aerobic exercise is performed on bicycle ergometers for a continuous 30 minutes with a progressive intensity of 40%-70% HRR. Resistance level is set according to an adaptive training prior to the first intervention, pedal cadences are 50-60r/min.

Resistance exercise is conducted using a set of equipment including chest press/ row, leg extension/ curl, abdominal/ back, biceps/ triceps, inner/ outer thigh, and push/ pull machines. Prior to conducting the 1 repetition maximum (RM) testing for the major muscles of the upper and lower limbs, all participants receive proper instructions on how to use the equipment. The Brzycki 1-RM prediction equation is used to estimate the 1RM based on the recorded resistance and repetitions. All participants performe resistance exercise with a weight of 60%-80% 1RM. Movements on each machine are repeated 10-12 times per unit for a total of 4 units, with a-30 second break between units.

In all intervention sessions, participants in AR group complete aerobic exercise before starting resistance exercise, while participants in RA group performe two types of exercise in a reversed order. Participants are instructed to maintain their usual lifestyle but refrain from engaging in other forms of regular exercise throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-70 years;
* Type 2 diabetes diagnosed as: random blood glucose ≥11.1mmol/L (200mg/dL) or fasting blood glucose ≥7.0mmol/L (126mg/L) or oral glucose tolerance test (2h) ≥11.1mmol/L (200mg/dL) or glycated hemoglobin (HbA1c) ≥ 6.5%;
* The course of type 2 diabetes lasted for one year or longer;
* Willing to participate and sign the informed consent form voluntarily

Exclusion Criteria:

* Type 1 diabetes;
* Fasting blood glucose (FBG)>16.7mmol/L;
* Severe complications of diabetes such as acute infection, diabetic ketoacidosis, and plantar lesions;
* Severe kidney disease, cardiovascular and cerebrovascular diseases as identified by a specialist;
* Musculoskeletal, neurological, psychiatric or other disorders which limit the ability to exercise as identified by a specialist;
* Doing physical exercise regularly (≥ 3 times per week, at least 1 hour per session of moderate to vigorous activities);
* Currently under dietary program for weight loss;
* Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg at rest;
* Abnormal electrocardiogram (rest and exercise);
* Other comorbidities or medications irrelevant to diabetes treatment that may influence glycemia during the past 6 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, MD, PhD, Study Director — Nanjing Sport Institute; Xiao Tan, PhD, Principal Investigator — Zhejiang University; Lijun Wei, MD, Study Director — Maigaoqiao Community Health Service Center
Locations (1):
- Maigaoqiao Community Health Service Center, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in outpatient clinics or via online/printed advertisement delivered through the Maigaoqiao Community Health Service Center from Oct 1st, 2023 to Nov 3rd, 2023.
Pre-assignment Details: The exclusion criteria included patients with T1D, diseases diagnosed by physicians that are unsuitable for exercise intervention, such as severe cardiovascular diseases, acute infections, musculoskeletal disorders, and other related conditions, patients who have regular physical activity habits (90min moderate intensity exercise or 75min high intensity exercise), and currently under dietary program for weight loss
Groups:
- AR Group: Aerobic Exercise Before Resistance Exercise: AR group: aerobic training before resistance training: Exercise are performed 3 times/wk for 8 wks.
  Aerobic training sessions are performed using cycle ergometers. Riding speed is 55-60 rotations/min, at an intensity between 50%-75% of heart rate reserve (HRR). Real-time heart rate monitors are worn by each participant during the session. Aerobic training session lasts for 30 minutes, with an additional 5-minute warm-up and 5-min relaxation training before and after the session, respectively.
  Participants perform resistance exercise on a set of strength training equipment. Load of resistance exercise is between 60-80% of repetition maximum (RM) in each set of exercise. Six different groups of resistance exercise (involving contractions and relaxations of biceps, triceps, pectoralis major, latissimus dorsi, quadriceps, and hamstrings) are conducted, with 6 sets of 10 repeated tasks in each group. Participants are instructed to finish each set of exercise task within 60 seconds. Between each two sets, there are 60 s of rest time.
- RA Group: Resistance Training Before Aerobic Training: RA group: resistance exercise before aerobic exercise: Exercise are performed 3 times/wk for 8 wks.
  Following a 5-min warm-up exercise, the participants perform resistance training on a set of equipment. Load of resistance exercise is set between 60-80% of repetition maximum in each set of exercise. Six different groups of resistance exercise (involving contractions and relaxations of biceps, triceps, pectoralis major, latissimus dorsi, quadriceps, and hamstrings) are conducted, with 6 sets of 10 repeated tasks in each group. Participants are instructed to finish each set of exercise task within 60 s. Between each two sets, there are 60 seconds of rest time.
  Aerobic training sessions are performed using cycle ergometers. Riding speed is 55-60 rotations/min, at an intensity between 50%-75% of heart rate reserve. Real-time heart rate monitors are worn during the entire session. Each aerobic training session lasts for 30 minutes, with an 5-minute relaxation training after the session.
Period: Overall Study
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (4.1) | 63.2 (4.5) | 62.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 12 | 14 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose at Baseline
Description: blood glucose level following overnight (12-h) fasting
Time Frame: At week 0, within 7 days before the intervention starts
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
mmol/L | 7.2 [6.7 to 8.2] | 7.0 [6.1 to 8.0]

2. Primary Outcome: Fasting Glucose at Follow-up
Description: blood glucose level following overnight (12-h) fasting
Time Frame: At week 9, within 7 days after the intervention completes
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
mmol/L | 7.2 [6.7 to 8.5] | 7.4 [6.2 to 8.2]

3. Primary Outcome: Hemoglobin A1c (HbA1c) at Baseline
Description: At baseline, the HbA1c level in blood among all participants
Time Frame: At baseline, within 7 days before the intervention starts
Measure: Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
percentage of glycated hemoglobin | 7.5 [6.8 to 8.2] | 7.3 [6.7 to 7.7]

4. Primary Outcome: Hemoglobin A1c (HbA1c) at Follow-up
Description: After intervention, the HbA1c level in blood among all participants
Time Frame: At week 9, within 7 days after the completion of the 8-week intervention
Measure: Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
percentage of glycated hemoglobin | 7.0 [6.8 to 7.7] | 7.2 [6.8 to 7.6]

5. Primary Outcome: Continuous Glucose Monitoring at Baseline (Mean, sd, Lage)
Description: At baseline, 14-day continuous glucose monitoring including mean, sd, cv, lage, tir, tar, tbr
Time Frame: At baseline, within 14 days before the intervention starts, measurement lasts for 14 days (mean, sd, lage)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
mmol/L
  mean glucose | 8.7 (1.3) | 8.1 (1.5)
  standard deviation of blood glucose | 2.2 (0.7) | 2.1 (0.6)
  largest amplitude of glucose excursion | 8.7 (1.9) | 8.3 (1.9)

6. Primary Outcome: Continuous Glucose Monitoring at Baseline (Coefficient of Variation)
Description: At baseline, 14-day continuous glucose monitoring including mean glucose value, standard deviation (SD) of the glucose values, coefficient of variation (CV) of relative standard deviation, LAGE, TIR, TAR, TBR
Time Frame: At baseline, within 14 days before the intervention starts, measurement lasts for 14 days (cv)
Measure: Mean (Standard Deviation); unit: % of relative standard deviation
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
% of relative standard deviation | 24.1 (5.6) | 25.1 (3.9)

7. Primary Outcome: Continuous Glucose Monitoring at Baseline (Tir, Tar, Tbr)
Description: At baseline, 14-day continuous glucose monitoring including mean, sd, cv, lage, tir, tar, tbr
Time Frame: At baseline, within 14 days before the intervention starts, measurement lasts for 14 days (tir, tar, tbr)
Measure: Mean (Standard Deviation); unit: % of measurement time
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
% of measurement time
  time in range | 72.3 (18.8) | 77.4 (16.7)
  time above range | 33.6 (26.4) | 23.9 (20.7)
  time below range | 0.4 (1.1) | 0.9 (2.1)

8. Primary Outcome: Continuous Glucose Monitoring at Follow-up (Mean, sd, Lage)
Description: After intervention, 14-day continuous glucose monitoring including mean, sd, cv, lage, tir, tar, tbr
Time Frame: at week 8-9
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
mmol/L
  Mean Glucose | 8.2 (1.0) | 8.4 (1.6)
  Standard Deviation of Blood Glucose | 2.4 (0.7) | 2.1 (0.5)
  Largest Amplitude of Glucose Excursion | 9.1 (2.2) | 8.1 (1.5)

9. Primary Outcome: Continuous Glucose Monitoring at Follow-up (Coefficient of Variation)
Description: as for outcome 6
Time Frame: at week 8-9
Measure: Mean (Standard Deviation); unit: % of relative standard deviation
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
% of relative standard deviation | 26.1 (4.4) | 25.6 (4.2)

10. Primary Outcome: Continuous Glucose Monitoring at Follow-up (Tir, Tar, Tbr)
Description: After intervention, 14-day continuous glucose monitoring including mean, sd, cv, lage, tir, tar, tbr
Time Frame: at week 8-9
Measure: Mean (Standard Deviation); unit: % of measurement time
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
Number analyzed (Participants) | 28 | 28
% of measurement time
  Time In Range | 75.9 (12.9) | 78.0 (13.9)
  Time Above Range | 27.6 (21.6) | 26.1 (20.6)
  Time Below Range | 1.4 (4.3) | 0.9 (2.1)

ADVERSE EVENTS:
Time Frame: Baseline assessments were implemented between November 7, 2023 and November 29, 2023. Intervention was performed between November 16, 2023 and January 21, 2024. Follow-up assessments were implemented between January 2, 2024 and February 2, 2024. Adverse event data were collected until July 2, 2024. For each participant, adverse event data was collected through approximately 8 months, which was from the first date of baseline assessments to 5 months after the end of follow-up assessments.
Arm/Group | AR Group: Aerobic Exercise Before Resistance Exercise | RA Group: Resistance Training Before Aerobic Training
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT06145542/Prot_SAP_000.pdf